CLINICAL TRIAL: NCT07168590
Title: The Effect of Radiographically Evaluated Anatomical Axis on Pain and Kinesiophobia in Knee Osteoarthritis
Brief Title: Anatomical Axis on X-Ray and Its Relationship With Pain and Kinesiophobia in Knee Osteoarthritis
Acronym: KOA-AXIS
Status: Not yet recruiting | Type: Observational
Sponsor: Selim Sezikli (Other Government)
Responsible Party: Sponsor-Investigator, Selim Sezikli, Medical Doctor, Specialist in Physical Medicine and Rehabilitation, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Organization: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Other Study IDs: KOA2025
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis; Pain; Kinesiophobia
Keywords: Knee osteoarthritis; Anatomical axis; Radiographic alignment; Tampa Scale for Kinesiophobia (TSK); SF-36; WOMAC; Pain; Femoro-tibial angle; Kinesiophobia
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee Osteoarthritis Patients: This cohort includes adult patients diagnosed with knee osteoarthritis who meet the inclusion criteria. All participants will undergo clinical evaluation of pain, functional status, quality of life, and kinesiophobia using validated scales (VAS, WOMAC, SF-36, TSK). Radiographic assessment will be performed on existing anteroposterior knee X-rays taken within the last 6 months, including femoro-tibial angle and joint space width measurements. No experimental intervention will be applied; data will be collected in an observational and cross-sectional manner.

SUMMARY:
Knee osteoarthritis is a common joint disease that causes pain, stiffness, and limitations in daily activities, especially in older adults. Changes in the alignment of the lower limb, called the anatomical axis, can increase the mechanical load on the knee joint and may affect pain and mobility. This study aims to investigate the relationship between the anatomical axis measured on knee X-rays and patients' pain levels, functional status, quality of life, and fear of movement (kinesiophobia).

This is a single-center, observational, cross-sectional study. Adult patients diagnosed with knee osteoarthritis who have a standard knee X-ray taken within the last 6 months and who volunteer to participate will be included. Pain will be measured with the Visual Analog Scale (VAS), functional status with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), quality of life with the 36-Item Short Form Health Survey (SF-36), and kinesiophobia with the Tampa Scale for Kinesiophobia (TSK). The femoro-tibial angle and joint space width will be measured on X-rays by two independent observers.

By examining the relationship between radiographic alignment and clinical findings, this study may provide new insights into the comprehensive evaluation of knee osteoarthritis and help guide treatment planning for patients.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a prevalent degenerative joint disease that leads to pain, disability, and reduced quality of life, particularly in older adults. Alterations in lower limb alignment, specifically deviations of the anatomical (mechanical) axis such as varus or valgus deformities, play a key role in the development and progression of OA by altering joint load distribution. Varus alignment is commonly associated with medial compartment OA, whereas valgus alignment is related to lateral compartment OA. Previous studies have reported that such malalignment may accelerate structural damage, increase pain, and contribute to functional impairment.

In addition to structural changes, chronic pain in OA patients can lead to fear of movement, known as kinesiophobia, which further limits physical activity and negatively affects functional outcomes. However, there are limited studies that simultaneously evaluate the relationship between radiographic alignment, pain, functional capacity, quality of life, and kinesiophobia.

This single-center, observational, cross-sectional study will be conducted at the outpatient Physical Medicine and Rehabilitation clinics of Istanbul Physical Medicine and Rehabilitation Training and Research Hospital. The target sample size is 100 patients with knee OA, based on a priori power analysis. Eligible participants must have an anteroposterior knee X-ray taken within the last six months. Pain intensity will be assessed with the Visual Analog Scale (VAS), functional status with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), quality of life with the Short Form-36 (SF-36), and kinesiophobia with the Tampa Scale for Kinesiophobia (TSK). Radiographic measurements, including femoro-tibial angle and joint space width, will be performed by two independent observers using standardized procedures.

Collected data will be analyzed using appropriate statistical methods. The findings are expected to provide a more comprehensive understanding of the relationship between anatomical axis alignment and clinical outcomes in knee OA. This may contribute to more effective treatment planning and patient management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis (clinical and radiographic)
* Having an anteroposterior knee X-ray taken within the last 6 months
* Voluntary agreement to participate in the study
* Cognitive ability sufficient to understand test instructions

Exclusion Criteria:

* History of knee surgery
* Illiteracy (inability to read/write)
* Refusal to participate
* Presence of orthopedic conditions that prevent walking (e.g., amputation, joint prosthesis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with knee osteoarthritis who are admitted to the Physical Medicine and Rehabilitation outpatient clinics of Istanbul Physical Medicine and Rehabilitation Training and Research Hospital. Participants must have a knee X-ray taken within the last 6 months and meet the study's eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-03-08 (Estimated)

PRIMARY OUTCOMES:
Pain Severity Assessed by Visual Analog Scale (VAS) | Day 1 (single assessment at baseline)
  Pain intensity during daily activities will be assessed using a 10-cm Visual Analog Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst imaginable pain.
Kinesiophobia Assessed by Tampa Scale for Kinesiophobia (TSK) | Day 1 (single assessment at baseline)
  Fear of movement will be measured with the Tampa Scale for Kinesiophobia (TSK), a validated questionnaire widely used in musculoskeletal conditions.

SECONDARY OUTCOMES:
Functional Status Assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Day 1 (single assessment at baseline)
  Functional status, stiffness, and pain will be assessed using the WOMAC index, a validated tool for patients with knee osteoarthritis.
Quality of Life Assessed by Short Form-36 (SF-36) | Day 1 (single assessment at baseline)
  General health-related quality of life will be evaluated using the SF-36, a standardized questionnaire covering physical, emotional, and social domains.
Radiographic Alignment Assessed by Femoro-Tibial Angle (FTA) | Day 1 (single assessment at baseline)
  The anatomical axis of the lower limb will be measured on standard anteroposterior knee radiographs by two independent observers.
Joint Space Width (JSW) on Knee X-Ray | Day 1 (single assessment at baseline)
  Medial and lateral joint space width will be measured on radiographs to evaluate structural severity of knee osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Sezikli, MD, Principal Investigator — Istanbul Physical Medicine and Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including demographic information, pain scores (VAS), functional outcomes (WOMAC), quality of life scores (SF-36), kinesiophobia scores (TSK), and radiographic measurements (femoro-tibial angle, joint space width), will be shared. Data will be made available upon reasonable request from qualified researchers with ethics committee approval and a signed data use agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data and supporting documents (protocol, SAP, ICF) will be available beginning 6 months after study completion (September 2026) and will remain available for up to 2 years (until March 2028).
Access Criteria: Qualified researchers with approval from an independent ethics committee and a signed data use agreement will be granted access to de-identified individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan, informed consent form). Data will be shared in anonymized format to ensure patient confidentiality. Access requests should be submitted to the principal investigator, and data will be provided electronically after approval.